CLINICAL TRIAL: NCT03857399
Title: An Open，Multicenter Clinic Trial of the Effectiveness，Safety and Pharmacokinetics in the Empiric Therapy of Patients With Persistent Fever and Agranulocytosis Using Local Caspofungin
Brief Title: Empiric Therapy of Patients With Persistent Fever and Agranulocytosis Using Caspofungin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cttq (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTTQ-CORE-101
Record Dates: First submitted 2018-11-16; First posted 2019-02-28 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2020-12

CONDITIONS: Fungal Infection
MeSH Terms: conditions — Mycoses | interventions — Caspofungin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm-1 (Experimental): Patients will be assigned to receive intravenous local caspofungin (70 mg on day 1 and 50 mg once daily),If the study therapy was well tolerated but fever persisted for four or more days and the patient's clinical condition deteriorated, the dosage could be increased to 70 mg once daily.For patients who have no evidence of baseline or breakthrough fungal infection, study therapy was administered until the absolute neutrophil count was at least 500 per cubic millimeter and for up to 72 hours thereafter. The onsite investigator determined the duration of therapy for patients with baseline or breakthrough fungal infections; however,it was recommended that treatment be given for at least 14 days and for at least 7 days after neutropenia and symptoms resolved.
  Interventions: Drug: Caspofungin
- Arm-2 (Active Comparator): Patients will be assigned to receive intravenous original caspofungin (70 mg on day 1 and 50 mg once daily),the therapeutical duration is 4 Days.
  Interventions: Drug: Caspofungin

INTERVENTIONS:
Drug: Caspofungin — Considering the possibility of fungal infection, we take empiric therapy for the patients with persistent fever and agranulocytosis using caspofungin for injection.
  Other Names: original caspofungin

SUMMARY:
The purpose of this study is evaluating the efficacy and safety of generics caspofungin in the treatment of the patients with neutropenic and fever.Another purpose of this study is comparing the pharmacokinetic characteristics of generics caspofungin and original medicine(Cancidas®) for providing a basis for clinical rational administration.

DETAILED DESCRIPTION:
Caspofungin, a member of the new echinocandin class of compounds，had been proved as effective as and generally better tolerated than liposomal amphotericin B when given as empirical antifungal therapy in patients with persistent fever and neutropenia，and It was approved by FDA in 2001.The generics caspofungin of Chia Tai TianQing Pharmaceutical Group Co. , Ltd. (CTTQ) will be approved by CFDA.The purpose of this study is evaluating the efficacy and safety of this generics caspofungin in the empirical antifungal therapy in patients with persistent fever and neutropenia.

This is a prospective,multicenter,randomized,controlled,open label study,the designed cases are 60 subjects.This study is divided into two stages,one is pharmacokinetics study stage ,the purpose of this stage is comparing the blood concentration of generics caspofungin and original medicine(Cancidas®) ,24 of 60 subjects will participate in this stage,the randomization in a 1:1 ratio will be performed at each group.The other 36 subjects will participate in another stage that is a single study,all subjects will use generics caspofungin.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years old
* The neutrophil counts of the patients with leukemia, lymphoma or other tumors undergoing chemotherapy or receiving hematopoietic stem cell transplantation are below 500 million/L for 96 hours at least,as well as the body temperatures are over 38.0 °C;
* It is ineffective using intravenous broad-spectrum antibacterial therapy lasting at least 96h;
* Estimated survival period > 3 months;
* Subjects voluntarily participate in the study and sign informed consent.

Exclusion Criteria:

* The subjects did not receive adequate antibacterial therapy;
* The subjects were received other antifungal medications within 14 days (except for fluconazole prophylaxis);
* It was confirmed or clinically diagnosed as invasive fungal infection;
* Subjects with liver dysfunction (ALT, AST exceeds the upper limit of normal value by 2 times);
* Subjects with renal insufficiency (Cr, BUN exceeds the upper limit of the normal value of 1.5 times);
* Subjects are allergic to the investigational product;
* Pregnant or lactating women;
* Simultaneous treatment with cyclosporine, tacrolimus, rifampicin, efavirenz, nevirapine, dexamethasone, phenytoin or carbamazepine;
* Other circumstances that investigators believe unsuitable for enrollment; （criteria 8 does not apply to Phase 2）

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-09-17 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Efficacy evaluation 7 days after drug withdrawal | 7 days after drug withdrawal
  Curative effect evaluation consists of five parts:The fever subsided during agranulocytosis; Breakthrough invasive fungal infections do not occur during or within 7 days after treatment; If any baseline invasive fungal infection is present, the therapy is effective; The patient was still alive when 7 days after drug withdrawal; The study was not terminated for drug-related toxicity or lacking of efficacy.
Peak Plasma Concentration (Cmax) | Day1,day3,day4 after the start of the dosing
  The peak plasma concentration after injection of caspofungin
Half-Life (t 1/2) | Day1 after the start of the dosing
  The time of duration from the starting of injection to half plasma concentration of caspofungin
Area under the plasma concentration versus time curve (AUC) | Day1,day3,day4 after the start of the study
  The area under the plasma concentration of caspofungin versus time curve from Day1 to Day4 after the fist dosing

SECONDARY OUTCOMES:
The duration of fever | 7 days after drug withdrawal
  The duration of the fever in patients
Survival rate | 7 days after drug withdrawal
  The number of surviving patients divided by the total number of patients

CONTACTS AND LOCATIONS:
Overall Officials: Jianda Hu, Ph.D, Principal Investigator — Affiliated Concord Hospital of Fujian Medical University
Locations (6):
- China (6):
  - Affiliated Concord Hospital of Fujian Medical University, Fuzhou, Fujian
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital of Suzhou University, Suzhou, Jiangsu
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Tongji Hospital of Shanghai, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang